CLINICAL TRIAL: NCT01659333
Title: Volume Status in Peritoneal Dialysis Patients With Using Different Determining Methods.
Brief Title: The Association Between Arterial Stiffness and Assessment of Hydration State in Peritoneal Dialysis Patients
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ismail Kocyigit, Associate Professor, TC Erciyes University
Other Study IDs: 2010/10
Record Dates: First submitted 2012-08-04; First posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Disorders Associated With Peritoneal Dialysis
Keywords: Peritoneal, Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Peritoneal dialysis, hypervolemia: All calculations are automatically performed by the software of the BCM device. Absolute over hydration (OH) is the difference between the expected patient's ECW under normal physiological conditions and the actual ECW, whereas the relative over hydration (Rel. OH) is defined as the OH to ECW ratio. Normohydration is defined when OH is between the 10th and the 90th percentile for healthy, age- and gender-matched individuals from the reference population, i.e., between 10th percentile (-1.1 L) to 90th percentile (+1.1 L), while volumes below and above this range define underhydration and overhydration, respectively.
- Peritoneal dialysis, normovolemia: All calculations are automatically performed by the software of the BCM device. Absolute over hydration (OH) is the difference between the expected patient's ECW under normal physiological conditions and the actual ECW, whereas the relative over hydration (Rel. OH) is defined as the OH to ECW ratio. Normohydration is defined when OH is between the 10th and the 90th percentile for healthy, age- and gender-matched individuals from the reference population, i.e., between 10th percentile (-1.1 L) to 90th percentile (+1.1 L), while volumes below and above this range define underhydration and overhydration, respectively.

SUMMARY:
Dry weight (DW) assessment is essential for the efficient treatment of peritoneal dialysis (PD) patients but so far objective methods for DW assessment have not been established for daily clinical practice. Our aim was to evaluate hydration state in PD patients by using a body composition monitor (BCM) and calf bioimpedance (c-BI) and N-terminal prohormone of brain natriuretic peptide (NT-proBNP) levels and to compare both methods with arterial stiffness.

DETAILED DESCRIPTION:
We evaluated 60 patients using a new BCM device that implies a validated body composition model. This method allows correct quantification of extracellular fluid overload or deficiency (normal limits:-1.1 to +1.1L). Patients were assigned to normo and hypervolemic groups according to BCM results. Also, normalized calf resistivity (nRho) was calculated from resistance at 5 Khz using c-BI and the levels of NT-proBNP were measured in all study patients. The analyses of arterial stiffness were performed by using the pulse wave velocity (PWV) technique on the patients. All patients underwent conventional echocardiography and their left ventricular diastolic functions were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal dialysis patients
* All participants over 18 years of age

Exclusion Criteria:

* Patients with valvular heart disease
* Patients with coronary artery disease
* Patients with cardiomyopathy
* Patients with ESRD who underwent hemodialysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We evaluated 60 patients' hydration states were measured by bioimpedance spectroscopy methods. Patients were assigned to normo and hypervolemic groups according to Body composition monitor(BCM) results. Also, normalized calf resistivity (nRho) was calculated from resistance at 5 Khz and the levels of NT-proBNP were measured in all study patients. The analyses of arterial stiffness were performed by using the pulse wave velocity (PWV) technique on the patients. Additionally, all patients underwent conventional echocardiography and their left ventricular diastolic functions were evaluated. The patients were grouped using the BCM method because, according to the literature, this method is the only one that can classify subjects in terms of volume conditions.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Terminated of patients recruiting | One year

CONTACTS AND LOCATIONS:
Overall Officials: Murat Sipahioglu, MD, Study Director — TC Erciyes University
Locations (1):
- Erciyes University Nephrology Department, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Kocyigit I, Sipahioglu MH, Orscelik O, Unal A, Celik A, Abbas SR, Zhu F, Tokgoz B, Dogan A, Oymak O, Kotanko P, Levin NW. The association between arterial stiffness and fluid status in peritoneal dialysis patients. Perit Dial Int. 2014 Nov-Dec;34(7):781-90. doi: 10.3747/pdi.2013.00057. Epub 2014 Jan 2. PMID 24385328
- See also: http://tip.erciyes.edu.tr/etikkurul_ana_sayfa.asp, more informaiton for our study in this link. — http://tip.erciyes.edu.tr/